CLINICAL TRIAL: NCT04598841
Title: A Multicentric Study on Pre-operative Nutritional Support for Hirschsprung's Disease
Brief Title: Nutrition Support for Hirschsprung Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Jiexiong Feng, professor, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: TJH-HSCRNS
Record Dates: First submitted 2020-10-18; First posted 2020-10-22 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: Nutrition Supporting; Hirschsprung Disease; Infants; Prospective Study
MeSH Terms: conditions — Hirschsprung Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): Intravenous nutrition or oral high-calorie diet 7-10 days before surgery
  Interventions: Dietary Supplement: supplement nutritional supporting
- control group (No Intervention): normal diet before surgery

INTERVENTIONS:
Dietary Supplement: supplement nutritional supporting — Special medical formula for the purpose of formula food
  Arms: intervention group

SUMMARY:
A multi-center, prospective,randomized, non-blind, controlled study was conducted to investigate the effects of different pre-operative nutritional support modes on perioperative nutritional status, surgical treatment success rate, and rehabilitation process in children with Hirschsprung disease.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 0-5 years.
2. Clinical diagnosis with Hirschsprung's disease who requires surgery;

Exclusion Criteria:

1. Complicated with severe complications such as enterocolitis associated with Hirschsprung disease;
2. History of diseases associated with various organ systems that may be life-threatening;
3. Other severe digestive tract malformations or other diseases that may interfere with the treatment or compliance of the child;
4. Patients who have participated in other clinical trials within the last 1 month;
5. Any other conditions in which the investigator considers it inappropriate to participate in the trial.

Ages: 0 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 110 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
rate of postoperative HAEC | 3 months
  Incidence of postoperative HAEC

SECONDARY OUTCOMES:
Z score | 3 months
  weight/age
LOS | 1 months
  length of postoperative stay
reoperation | 3 months
  rate of reoperation
readmission | 3 months
  rate of readmission

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

REFERENCES:
- [Derived] Zhang HY, Chen K, Zhang Y, Gao T, Huang Y, Ge L, Yuan Y, Zhang G, Yang H, Ren H, Zhan J, Xu W, Liu X, Zhu T, Feng J. Preoperative nutritional support in children with Hirschsprung disease: a prospective multicenter open-label randomized controlled trial. Nat Commun. 2025 Dec 19;16(1):11171. doi: 10.1038/s41467-025-66541-x. PMID 41419466